CLINICAL TRIAL: NCT00395512
Title: A Multicenter, Double-Blind Study to Determine the Efficacy and Safety of SYR-322 Plus Pioglitazone HCl (Actos®), SYR-322 Alone or Pioglitazone HCl Alone in Subjects With Type 2 Diabetes
Brief Title: Efficacy of Alogliptin With Pioglitazone (Actos®) in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-06-TL-322OPI-002; 2006-005492-17 (EudraCT Number); U1111-1113-8616 (Registry Identifier: WHO)
Record Dates: First submitted 2006-11-01; First posted 2006-11-03 (Estimated); Results first posted 2013-03-27 (Estimated); Last update posted 2013-03-27 (Estimated); Status verified 2013-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — alogliptin; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Alogliptin 25 mg QD (Experimental): Alogliptin 25 mg, tablets, orally, once daily and pioglitazone placebo-matching tablets, orally, once daily for up to 26 weeks.
  Interventions: Drug: Alogliptin; Drug: Placebo
- Pioglitazone 30 mg QD (Active Comparator): Pioglitazone 30 mg, tablets, orally, once daily and alogliptin placebo-matching tablets, orally, once daily for up to 26 weeks.
  Interventions: Drug: Pioglitazone; Drug: Placebo
- Alogliptin 25 mg QD+ Pioglitazone 30 mg QD (Experimental): Alogliptin 25 mg, tablets, orally, once daily and pioglitazone 30 mg, tablets, orally, once daily for up to 26 weeks.
  Interventions: Drug: Alogliptin; Drug: Pioglitazone
- Alogliptin 12.5 mg QD + Pioglitazone 30 mg QD (Active Comparator): Alogliptin 12.5 mg, tablets, orally, once daily and pioglitazone 30 mg, tablets, orally, once daily for up to 26 weeks.
  Interventions: Drug: Alogliptin; Drug: Pioglitazone

INTERVENTIONS:
Drug: Alogliptin — Alogliptin tablets.
  Other Names: SYR-322
  Arms: Alogliptin 12.5 mg QD + Pioglitazone 30 mg QD; Alogliptin 25 mg QD; Alogliptin 25 mg QD+ Pioglitazone 30 mg QD
Drug: Pioglitazone — Pioglitazone tablets.
  Other Names: Actos; AD4833
  Arms: Alogliptin 12.5 mg QD + Pioglitazone 30 mg QD; Alogliptin 25 mg QD+ Pioglitazone 30 mg QD; Pioglitazone 30 mg QD
Drug: Placebo — Matching placebo tablets.
  Arms: Alogliptin 25 mg QD; Pioglitazone 30 mg QD

SUMMARY:
The purpose of this study is to evaluate the combination of alogliptin, once daily (QD), and pioglitazone in patients with type 2 diabetes mellitus who are inadequately controlled with diet and exercise alone.

DETAILED DESCRIPTION:
There are approximately 19 million people in the United States who have been diagnosed with diabetes mellitus, of which 90% to 95% is type 2. The prevalence of type 2 diabetes varies among racial and ethnic populations and has been shown to correlate with age, obesity, family history, history of gestational diabetes, and physical inactivity. Over the next decade, a marked increase in the number of adults with diabetes mellitus is expected, placing an ever-increasing burden on families and the health care system.

Current pharmacologic interventions for type 2 diabetes mellitus include a diverse range of antidiabetic medications with different mechanisms of action including insulin and insulin analogues, sulfonylureas, metformin, meglitinides, thiazolidinediones, inhibitors of alpha- glucosidase, analogs of glucagon-like peptide-1, and synthetic analogues of human amylin. Despite the variety of medications, many have clinically important or potentially life-threatening side effects, restricted use in many subpopulations, concerns with long-term tolerability, and challenges related to compliance due to side effects and route of administration. All of these reasons contribute to the difficulties patients have reaching the target glycosylated hemoglobin level less than 7%.

SYR-322 (alogliptin) is a selective, orally available inhibitor of the dipeptidyl peptidase-4 enzyme. Dipeptidyl peptidase-4 enzyme is thought to be primarily responsible for the in vivo degradation of 2 peptide hormones released in response to nutrient ingestion, namely glucagon-like peptide-1 and glucose-dependent insulinotropic peptide. Both peptides exert important effects on islet beta cells to stimulate glucose-dependent insulin secretion as well as regulating beta cell proliferation and cytoprotection. Glucagon-like peptide-1, but not glucose-dependent insulinotropic peptide, inhibits gastric emptying, glucagon secretion, and food intake. Glucose-dependent insulinotropic peptide has been shown to enhance insulin secretion by direct interaction with a glucose-dependent insulinotropic peptide -specific receptor on islet beta cells. The glucose-lowering actions of glucagon-like peptide-1, but not glucose-dependent insulinotropic peptide, are preserved in patients with type 2 diabetes mellitus.

Pioglitazone (ACTOS®) is a thiazolidinedione developed by Takeda Chemical Industries, Ltd. (Osaka, Japan) that is approved for the treatment of type 2 diabetes mellitus. Pioglitazone is a selective peroxisome proliferator-activated receptor-gamma agonist that decreases insulin resistance in the periphery and liver resulting in increased insulin-dependent glucose disposal and decreased hepatic glucose output.

As the rate of newly diagnosed cases of type 2 diabetes mellitus continues to grow, so does the need for products that will provide better glycemic control and improved safety and tolerability. Alogliptin and pioglitazone have complementary actions. Alogliptin inhibits the degradation of glucagon-like peptide-1 by inhibiting the enzyme dipeptidyl peptidase IV, thus augmenting glucose-dependent insulin secretion while pioglitazone is a peripheral and hepatic insulin sensitizer. Given the complementary mechanisms of action of alogliptin (stimulates insulin secretion) and pioglitazone (enhances insulin sensitivity), the addition of combination therapy in treatment naïve type 2 diabetes patients may potentially allow the patients to reach and maintain their glycosylated hemoglobin goal more effectively.

The aim of this study is to evaluate the effectiveness of the combination of alogliptin with pioglitazone in patients who are inadequately controlled on diet and exercise alone. Study participation is anticipated to be approximately 8.5 months.

ELIGIBILITY:
Inclusion Criteria

* Historical diagnosis of type 2 diabetes.
* Failed treatment with diet and exercise for at least 2 months prior to Screening.
* Is experiencing inadequate glycemic control as defined as glycosylated hemoglobin concentration between 7.5-11%, inclusive.
* Has received any antidiabetic therapy for less than 7 days within 3 months prior to Screening.
* Has a body mass index greater than or equal to 23 kg/m2 and less than or equal to45 kg/m2.
* Fasting C-peptide greater than or equal to 0.8 ng per mL.
* Regular use of other, non-excluded medications is allowed if participant is on a stable dose for at least 4 weeks prior to Screening.
* Females of childbearing potential who are sexually active must agree to use adequate contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Must be willing and able to monitor their blood concentrations with a home glucose monitor.

Exclusion Criteria

* Systolic blood pressure greater than or equal to 160 mmHg and diastolic blood pressure greater than or equal to 100 mmHg.
* Hemoglobin less than or equal to 12 g per dL for males and less than or equal to 10 g per dL for females.
* Alanine aminotransferase greater than or equal to 2.5times the upper limit of normal.
* Serum creatinine greater than 2.0 mg per dL.
* Thyroid stimulating hormone level greater than the upper limit of normal range.
* Major illness or debility that in the investigator's opinion prohibits the subject from completing the study.
* Urine albumin to creatinine ratio of greater than 1000 ug per mg at Screening. If elevated, the subject may be rescreened within 1 week.
* History of cancer, other than squamous cell or basal cell carcinoma of the skin, that has not been in full remission for at least 5 years prior to Screening
* History of laser treatment for proliferative diabetic retinopathy within 6 months prior to Screening.
* History of gastroparesis.
* Has New York Heart Association Class I to IV heart failure regardless of therapy.
* History of coronary angioplasty, coronary stent placement, coronary bypass surgery, or myocardial infarction within 6 months prior to Screening.
* History of any hemoglobinopathy that may affect determination of glycosylated hemoglobin.
* History of infection with hepatitis B, hepatitis C, or human immunodeficiency virus.
* History of a psychiatric disorder that will affect participant's ability to participate in the study.
* History of angioedema in association with use of angiotensin-converting enzyme inhibitors or angiotensin-II receptor inhibitors.
* Any alteration in angiotensin-II receptor inhibitors within 2 months prior to Randomization, if applicable.
* History of alcohol (defined as regular or daily consumption of more than 4 alcoholic drinks per day) or substance abuse (defined as illicit drug use) within 2 years prior to Screening.
* Received any investigational drug within 30 days prior to Screening or a history of receipt of an investigational antidiabetic drug within 3 months prior to Screening.
* Previously participated in an investigational study of SYR-322.
* Glycosylated hemoglobin concentration between 7.5-11%, inclusive, and a fasting plasma glucose less than 310 mg per dL.
* At least 75% compliant with the single-blind placebo regimen during the run-in/stabilization period.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 655 (Actual)
Dates: Start 2006-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP, Biological Sciences, Study Director — Takeda
Locations (161):
- United States (83):
  - Columbiana, Alabama
  - Hueytown, Alabama
  - Huntsville, Alabama
  - Northport, Alabama
  - Tucson, Arizona
  - Jonesboro, Arkansas
  - Little Rock, Arkansas
  - Searcy, Arkansas
  - Foothill Ranch, California
  - Irvine, California
  - Northridge, California
  - San Diego, California
  - San Mateo, California
  - Santa Monica, California
  - Jacksonville, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Port Charlotte, Florida
  - Sebastian, Florida
  - South Miami, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - Barnesville, Georgia
  - Columbus, Georgia
  - Savannah, Georgia
  - Chicago, Illinois
  - Libertyville, Illinois
  - South Bend, Indiana
  - Bossier City, Louisiana
  - Elkton, Maryland
  - Prince Frederick, Maryland
  - Towson, Maryland
  - North Dartmouth, Massachusetts
  - Bay City, Michigan
  - Benzonia, Michigan
  - Portage, Michigan
  - Saint Clair Shores, Michigan
  - Picayune, Mississippi
  - St Louis, Missouri
  - Billings, Montana
  - Las Vegas, Nevada
  - Elizabeth, New Jersey
  - Hamilton, New Jersey
  - Cicero, New York
  - Charlotte, North Carolina
  - Mooresville, North Carolina
  - Northeast, North Dakota
  - Franklin, Ohio
  - Ashland, Oregon
  - Altoona, Pennsylvania
  - Fleetwood, Pennsylvania
  - Harleysville, Pennsylvania
  - Havertown, Pennsylvania
  - Norristown, Pennsylvania
  - Northern Cambria, Pennsylvania
  - Penndel, Pennsylvania
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Florence, South Carolina
  - Orangeburg, South Carolina
  - Taylors, South Carolina
  - Williamston, South Carolina
  - Morristown, Tennessee
  - Arlington, Texas
  - Colleyville, Texas
  - Conroe, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Euless, Texas
  - Fort Worth, Texas
  - Garland, Texas
  - Houston, Texas
  - Katy, Texas
  - San Antonio, Texas
  - Seguin, Texas
  - Sugarland, Texas
  - Tomball, Texas
  - Ogden, Utah
  - Arlington, Virginia
  - Norfolk, Virginia
  - Richmond, Virginia
  - Lewisburg, West Virginia
  - Milwaukee, Wisconsin
- Argentina (6):
  - Cap. Fed., Buenos Aires
  - Chacabuco, Buenos Aires
  - La Plata, Buenos Aires
  - Mar del Plata, Buenos Aires
  - Morón, Buenos Aires
  - Córdoba
- Australia (3):
  - Kingswood, New South Wales
  - Fitzroy, Victoria
  - Frankston, Victoria
- Brazil (7):
  - Fortaleza, Ceará
  - Goiás, Goiás
  - Curitiba, Paraná
  - Belém, Pará
  - Maringá, RP
  - Marília, São Paulo
  - Mogi das Cruzes, São Paulo
- Pleven, Bulgaria
- Santiago, Chile
- Slavonski Brod, Croatia
- Pärnu, Estonia
- Guatemala City, Guatemala
- Hungary (6):
  - Budapest
  - Eger
  - Gyula
  - Makó
  - Nyíregyháza
  - Pécs
- India (6):
  - Hyderabad, Andhra Pradesh
  - Bangalore, Karnataka
  - Aurangabad, Maharashtra
  - Mumbai, Maharashtra
  - Nagpur, Maharashtra
  - Chennai, Tamil Nadu
- Israel (6):
  - Hadera
  - Haifa
  - Holon
  - Jaffa Tel Aviv
  - Jerusalem
  - Nahariya
- Riga, Latvia
- Lithuania (2):
  - Kaunas
  - Kėdainiai
- Mexico (3):
  - Aguascalientes
  - Mexico City
  - Monterrey
- New Zealand (2):
  - Christchurch
  - Hamilton
- Poland (7):
  - Bialystok
  - Bytom
  - Gdansk
  - Gniewkowo
  - Kamieniec Ząbkowicki
  - Krakow
  - Łęczyca
- Romania (3):
  - Brasov
  - Bucharest
  - Galati
- Russia (3):
  - Kazan'
  - Moscow
  - Yekaterinburg
- Serbia (3):
  - Belgrade
  - Kragujevac
  - Niš
- Slovakia (5):
  - Interna Klinika II, Nitra Region
  - Banska Bysterica
  - Lučenec
  - Riverside
  - Šahy
- South Africa (6):
  - Port Elizabeth, Eastern Cape
  - Johannesburg, Gauteng
  - Durban, KwaZulu-Natal
  - East Lynne, Pretoria
  - Bellville, Western Province
  - Cape Town, Western Province
- Ukraine (4):
  - Dnipropetrovsk
  - Kharkiv
  - Lviv
  - Odesa

REFERENCES:
- [Result] Rosenstock J, Inzucchi SE, Seufert J, Fleck PR, Wilson CA, Mekki Q. Initial combination therapy with alogliptin and pioglitazone in drug-naive patients with type 2 diabetes. Diabetes Care. 2010 Nov;33(11):2406-8. doi: 10.2337/dc10-0159. Epub 2010 Aug 19. PMID 20724648
- See also: ACTOS® Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ACTOSPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 268 investigative sites in 23 countries from 02 November 2006 to 13 February 2008.
Pre-assignment Details: Participants with a diagnosis of type 2 diabetes who were inadequately controlled with diet and exercise were randomized to 1 of 4 treatment groups in a 1:1:1:1 ratio as follows: Alogliptin alone, pioglitazone alone, alogliptin 25 mg + pioglitazone 30 mg and alogliptin 12.5 mg + pioglitazone 30 mg.
Groups:
- Alogliptin 25 mg: Alogliptin 25 mg, tablets, orally, once daily and pioglitazone placebo-matching tablets, orally, once daily for up to 26 weeks.
- Pioglitazone 30 mg: Pioglitazone 30 mg, tablets, orally, once daily and alogliptin placebo-matching tablets, orally, once daily for up to 26 weeks.
- Alogliptin 25 mg + Pioglitazone 30 mg: Alogliptin 25 mg, tablets, orally, once daily and pioglitazone 30 mg, tablets, orally, once daily for up to 26 weeks.
- Alogliptin 12.5 mg + Pioglitazone 30 mg: Alogliptin 12.5 mg, tablets, orally, once daily and pioglitazone 30 mg, tablets, orally, once daily for up to 26 weeks.
Period: Overall Study
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Started | 164 | 163 | 164 | 164
Safety Set | 164 | 163 | 164 | 163 (1 participant was lost to follow-up post visit 1. It is unknown if they took any study medication.)
Completed | 126 | 126 | 136 | 126
Not Completed | 38 | 37 | 28 | 38
Not completed — Adverse Event | 3 | 8 | 6 | 6
Not completed — Protocol Violation | 2 | 3 | 6 | 7
Not completed — Lost to Follow-up | 2 | 6 | 5 | 5
Not completed — Withdrawal by Subject | 6 | 5 | 5 | 12
Not completed — Physician Decision | 6 | 4 | 2 | 2
Not completed — Other | 1 | 1 | 0 | 0
Not completed — Hyperglycemic Rescue | 18 | 10 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg | Total
Number analyzed (Participants) | 164 | 163 | 164 | 164 | 655
Age Continuous [Mean (Standard Deviation); unit: years] | 52.6 (10.38) | 51.5 (10.72) | 52.8 (11.01) | 53.5 (11.37) | 52.6 (10.88)
Age, Customized [Number; unit: participants]
  < 65 years | 144 | 143 | 140 | 130 | 557
  ≥ 65 years | 20 | 20 | 24 | 34 | 98
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 73 | 91 | 83 | 335
  Male | 76 | 90 | 73 | 81 | 320
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 63 | 65 | 58 | 62 | 248
  Not Hispanic or Latino | 101 | 98 | 106 | 102 | 407
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 14 | 15 | 12 | 16 | 57
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 8 | 9 | 12 | 9 | 38
  White | 135 | 130 | 129 | 132 | 526
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 9 | 11 | 6 | 32
Weight [Mean (Standard Deviation); unit: kg] | 86.72 (19.033) | 85.53 (16.254) | 85.39 (20.374) | 84.38 (20.378) | 85.50 (19.062)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 31.61 (5.587) | 30.87 (4.938) | 31.32 (5.354) | 30.71 (5.621) | 31.13 (5.382)
Duration of diabetes [Mean (Standard Deviation); unit: years] | 3.23 (3.559) | 3.20 (3.739) | 3.05 (3.328) | 3.36 (4.166) | 3.21 (3.704)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 26 in Glycosylated Hemoglobin (HbA1c)
Description: The change from Baseline to Week 26 in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound).
Time Frame: Baseline and Week 26
Population: The Full analysis Set (all randomized patients who took at least 1 dose of double-blind study drug) where a Baseline and at least 1 postbaseline value were available. Last observation carried forward (LOCF) imputation was utilized.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 160 | 153 | 158 | 158
percentage of glycosylated hemoglobin | -0.96 (0.081) | -1.15 (0.083) | -1.71 (0.081) | -1.56 (0.081)
Statistical Analysis 1: Comparison: Pioglitazone 30 mg vs Alogliptin 25 mg + Pioglitazone 30 mg; The primary efficacy variable was defined as change from Baseline in HbA1c level at Week 26. The null hypothesis was that the average change from Baseline in HbA1c at Week 26 for the A25 + P30 group would be equal to the average changes for the P30 alone and A25 alone groups; further, under the null hypothesis, the average change from Baseline in HbA1c at Week 26 for the A12.5 + P30 group was equal to the average change for the P30 alone group; Test type: Superiority or Other; p < 0.001, ANCOVA — ANCOVA model with treatment and geographic region as class variables and baseline HbA1c as a covariate; LS Mean Difference = -0.56, 95% CI 2-sided [-0.78 to -0.33]
Statistical Analysis 2: Comparison: Alogliptin 25 mg vs Alogliptin 25 mg + Pioglitazone 30 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — ANCOVA model with treatment and geographic region as class variables and baseline HbA1c as a covariate; LS Mean Difference = -0.75, 95% CI 2-sided [-0.98 to -0.53]
Statistical Analysis 3: Comparison: Pioglitazone 30 mg vs Alogliptin 12.5 mg + Pioglitazone 30 mg; Test type: Superiority or Other; p < 0.001, ANCOVA — ANCOVA model with treatment and geographic region as class variables and baseline HbA1c as a covariate; LS Mean Difference = -0.40, 95% CI 2-sided [-0.63 to -0.18]

2. Secondary Outcome: Change From Baseline in HbA1c Over Time
Description: The change from Baseline in HbA1c (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) at 4 week intervals during the study. Least Squares Means were from an Analysis of Covariance (ANCOVA) model with treatment and geographic region as class variables and baseline HbA1c as a covariate.
Time Frame: Baseline and Weeks 4, 8, 12, 16 and 20.
Population: The full analysis set where Baseline and at least 1 postbaseline value were available. Last observation carried forward (LOCF) imputation was utilized.
Measure: Least Squares Mean (Standard Error); unit: percentage of glycosylated hemoglobin
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
percentage of glycosylated hemoglobin
  Week 4 (n=145, 146, 144, 150) | -0.55 (0.043) | -0.30 (0.043) | -0.62 (0.043) | -0.51 (0.043)
  Week 8 (n=160, 153, 158, 158) | -0.84 (0.058) | -0.72 (0.060) | -1.19 (0.059) | -1.03 (0.059)
  Week 12 (n=160, 153, 158, 158) | -0.98 (0.070) | -1.04 (0.071) | -1.57 (0.070) | -1.34 (0.070)
  Week 16 (n=160, 153, 158, 158) | -1.01 (0.080) | -1.17 (0.082) | -1.67 (0.081) | -1.43 (0.081)
  Week 20 (n=160, 153, 158, 158) | -1.00 (0.077) | -1.20 (0.079) | -1.72 (0.078) | -1.54 (0.078)
Statistical Analysis 1: Comparison: Pioglitazone 30 mg vs Alogliptin 12.5 mg + Pioglitazone 30 mg; Comparison of change from Baseline at Week 20 between Pioglitazone 30 mg and Alogliptin 12.5 mg + Pioglitazone 30 mg; Test type: Superiority or Other; p = 0.003, ANCOVA; ANCOVA model with treatment and geographic region as class variables and baseline HbA1c as a covariate; LS Mean Difference = -0.33, 95% CI 2-sided [-0.55 to -0.12]
Statistical Analysis 2: Comparison: Pioglitazone 30 mg vs Alogliptin 25 mg + Pioglitazone 30 mg; Comparison of change from Baseline at Week 20 between Pioglitazone 30 mg and Alogliptin 25 mg + Pioglitazone 30 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model with treatment and geographic region as class variables and baseline HbA1c as a covariate; LS Mean Difference = -0.52, 95% CI 2-sided [-0.74 to -0.30]
Statistical Analysis 3: Comparison: Alogliptin 25 mg vs Alogliptin 25 mg + Pioglitazone 30 mg; Comparison of change from Baseline at Week 20 between Alogliptin 25 mg and Alogliptin 25 mg + Pioglitazone 30 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model with treatment and geographic region as class variables and baseline HbA1c as a covariate; LS Mean Difference = -0.73, 95% CI 2-sided [-0.94 to -0.51]

3. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose Over Time
Description: The change from Baseline in fasting plasma glucose was assessed at weeks 1, 2, 4, 8, 12, 16, 20 and 26. Least Squares Means were from an ANCOVA model with treatment and geographic region as class variables and baseline plasma glucose as a covariate.
Time Frame: Baseline and Weeks 1, 2, 4, 8, 12, 16, 20 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
mg/dL
  Week 1 (n=148, 146, 152, 151) | -14.6 (2.93) | -7.3 (2.95) | -26.6 (2.90) | -23.3 (2.91)
  Week 2 (n=161, 156, 162, 159) | -16.7 (2.87) | -14.2 (2.92) | -33.5 (2.87) | -30.9 (2.90)
  Week 4 (n=162, 157, 162, 161) | -26.7 (2.72) | -31.9 (2.76) | -41.4 (2.72) | -39.7 (2.73)
  Week 8 (n=162, 157, 162, 162) | -29.0 (2.80) | -38.0 (2.84) | -50.4 (2.80) | -48.4 (2.81)
  Week 12 (n=162, 157, 162, 162) | -29.5 (3.01) | -42.4 (3.05) | -51.9 (3.01) | -49.3 (3.01)
  Week 16 (n=162, 157, 162, 162) | -26.9 (3.11) | -40.6 (3.16) | -52.7 (3.12) | -46.6 (3.12)
  Week 20 (n=162, 157, 162, 162) | -28.3 (3.06) | -42.0 (3.11) | -54.0 (3.07) | -47.5 (3.07)
  Week 26 (n=162, 157, 162, 162) | -25.8 (3.26) | -37.3 (3.31) | -50.2 (3.27) | -48.5 (3.27)
Statistical Analysis 1: Comparison: Pioglitazone 30 mg vs Alogliptin 12.5 mg + Pioglitazone 30 mg; Comparison of change from Baseline in fasting plasma glucose at Week 26 between Pioglitazone 30 mg and Alogliptin 12.5 mg + Pioglitazone 30 mg; Test type: Superiority or Other; p = 0.017, ANCOVA; P-value is from an ANCOVA model with treatment and geographic region as class variables and Baseline fasting plasma glucose as covariate; LS Mean Difference = -11.2, 95% CI 2-sided [-20.3 to -2.0]
Statistical Analysis 2: Comparison: Pioglitazone 30 mg vs Alogliptin 25 mg + Pioglitazone 30 mg; Comparison of change from Baseline in fasting plasma glucose at Week 26 between Pioglitazone 30 mg and Alogliptin 25 mg + Pioglitazone 30 mg; Test type: Superiority or Other; p = 0.006, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -12.9, 95% CI 2-sided [-22.0 to -3.8]
Statistical Analysis 3: Comparison: Alogliptin 25 mg vs Alogliptin 25 mg + Pioglitazone 30 mg; Comparison of change from Baseline in fasting plasma glucose at Week 26 between Alogliptin 25 mg and Alogliptin 25 mg + Pioglitazone 30 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference = -24.5, 95% CI 2-sided [-33.5 to -15.4]

4. Secondary Outcome: Percentage of Participants With Marked Hyperglycemia
Description: Marked Hyperglycemia is defined as fasting plasma glucose greater than or equal to 200 mg/dL. Study week windows are defined to place hyperglycemia into visit categories.
Time Frame: Weeks 1, 2, 4, 8, 12, 16, 20 and 26.
Population: Full analysis set including patients with at least one non-missing fasting plasma glucose result in the specified interval in each treatment group.
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
percentage of participants
  Week 1 to < Week 4 (n=162, 157, 162, 161) | 31.5 | 31.8 | 18.5 | 28.6
  Week 4 to < Week 8 (n=153, 147, 148, 147) | 19.0 | 15.0 | 10.8 | 14.3
  Week 8 to < Week 12 (n=151, 146, 152, 146) | 15.2 | 11.6 | 7.2 | 8.2
  Week 12 to < Week 16 (n=153, 141, 148, 139) | 16.3 | 9.2 | 8.1 | 7.9
  Week 16 to < Week 20 (n=142, 135, 144, 131) | 16.2 | 14.8 | 2.8 | 6.9
  Week 20 to Week 26 (n=130, 132, 143, 128) | 17.7 | 11.4 | 10.5 | 6.3
  Overall (n=162, 157, 162, 162) | 44.4 | 38.2 | 25.3 | 30.9

5. Secondary Outcome: Percentage of Participants Meeting Rescue Criteria
Description: Rescue was defined as meeting 1 of the following criteria, confirmed by a 2nd sample drawn within 5 days after the first sample and analyzed by the central laboratory:
  1. After more than 4 weeks of treatment but prior to the Week 8 Visit: a single fasting plasma glucose ≥310 mg/dL (≥17.5 mmol/L);
  2. From the Week 8 Visit but prior to the Week 12 Visit: a single fasting plasma glucose ≥275 mg/dL (≥15.27 mmol/L);
  3. From the Week 12 Visit through the End-of-Treatment Visit: HbA1c ≥8.5% and ≤0.5% reduction in HbA1c as compared with the Baseline HbA1c.
Time Frame: Weeks 4, 8, 12, 16, 20 and 26.
Population: Full analysis set including patients with visits during or after the specified interval in each treatment group.
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
percentage of participants
  Week 4 to < Week 8 (n=160, 156, 161, 160) | 0 | 0 | 0 | 0.6
  Week 8 to < Week 12 (n=158, 151, 157, 153) | 1.3 | 0 | 0 | 0
  Week 12 to < Week 16 (n=156, 145, 153, 144) | 2.6 | 3.4 | 1.3 | 2.1
  Week 16 to < Week 20 (n=150, 138, 149, 134) | 7.3 | 2.2 | 0 | 1.5
  Week 20 to Week 26 (n=132, 133, 146, 130) | 0.8 | 1.5 | 1.4 | 0
  Overall (n=160, 156, 161, 160) | 11.3 | 6.4 | 2.5 | 3.8

6. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin Less Than or Equal to 6.5%
Description: Clinical response at Week 26 was assessed by the percentage of participants with HbA1c ≤6.5%.
Time Frame: Week 26
Population: Full Analysis Set. Participants who did not complete the scheduled Week 26 visit were assessed based on their response at the time of discontinuation.
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
percentage of participants | 11.6 | 16.6 | 27.4 | 26.4

7. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin Less Than or Equal to 7.0%
Description: Clinical response at Week 26 was assessed by the percentage of participants with HbA1c ≤ 7%.
Time Frame: Week 26
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
percentage of participants | 24.4 | 33.7 | 62.8 | 53.4

8. Secondary Outcome: Percentage of Participants With Glycosylated Hemoglobin Less Than or Equal to 7.5%
Description: Clinical response at Week 26 was assessed by the percentage of participants with HbA1c ≤ 7.5%.
Time Frame: Week 26
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
percentage of participants | 44.5 | 55.8 | 72.0 | 72.4

9. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin Greater Than or Equal to 0.5%
Description: Clinical response at Week 26 was assessed by the percentage of participants with a decrease from Baseline in HbA1c of ≥ 0.5%.
Time Frame: Baseline and Week 26
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
percentage of participants | 66.5 | 70.6 | 89.6 | 85.3

10. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin Greater Than or Equal to 1.0%
Description: Clinical response at Week 26 was assessed by the percentage of participants with a decrease from Baseline in HbA1c of ≥ 1%.
Time Frame: Baseline and Week 26
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
percentage of participants | 43.3 | 54.6 | 75.6 | 68.1

11. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin Greater Than or Equal to 1.5%.
Description: Clinical response at Week 26 was assessed by the percentage of participants with a decrease from Baseline in HbA1c of ≥ 1.5%.
Time Frame: Baseline and Week 26
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
percentage of participants | 29.3 | 33.1 | 57.3 | 50.9

12. Secondary Outcome: Percentage of Participants With a Decrease in Glycosylated Hemoglobin Greater Than or Equal to 2.0%
Description: Clinical response at Week 26 was assessed by the percentage of participants with a decrease from Baseline in HbA1c of ≥ 2.0%.
Time Frame: Baseline and Week 26
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
percentage of participants | 17.7 | 19.6 | 34.1 | 33.1

13. Secondary Outcome: Change From Baseline in Fasting Proinsulin
Description: Proinsulin is a precursor to insulin, and was measured as an indicator of pancreatic function. The change from Baseline in fasting proinsulin was assessed at Weeks 4, 8, 12, 16, 20 and 26. Least Squares Means were from an ANCOVA model with treatment and geographic region as class variables and baseline proinsulin as a covariate.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: pmol/L
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
pmol/L
  Week 4 (n=136, 134, 135, 145) | -4.9 (1.74) | -12.1 (1.75) | -16.0 (1.74) | -12.3 (1.68)
  Week 8 (n=150, 143, 146, 155) | -3.7 (1.57) | -14.9 (1.60) | -18.2 (1.59) | -17.7 (1.54)
  Week 12 (n=150, 143, 147, 155) | -5.9 (1.48) | -16.0 (1.52) | -18.6 (1.50) | -16.7 (1.46)
  Week 16 (n=150, 143, 147, 155) | -3.4 (1.88) | -16.3 (1.93) | -16.0 (1.90) | -13.1 (1.85)
  Week 20 (n=150, 143, 147, 155) | -8.1 (1.75) | -16.1 (1.79) | -19.8 (1.76) | -15.5 (1.72)
  Week 26 (n=150, 143, 147, 155) | -4.8 (1.64) | -13.2 (1.68) | -18.3 (1.66) | -15.1 (1.61)

14. Secondary Outcome: Change From Baseline in Insulin
Description: The change from Baseline in fasting insulin was assessed at Weeks 4, 8, 12, 16, 20 and 26. Least Squares Means were from an ANCOVA model with treatment and geographic region as class variables and baseline insulin as a covariate.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: μIU/mL
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
μIU/mL
  Week 4 (n=135, 133, 133, 145) | 0.43 (0.684) | -4.74 (0.689) | -4.67 (0.687) | -4.27 (0.659)
  Week 8 (n=150, 142, 147, 155) | 0.93 (0.811) | -4.41 (0.834) | -4.75 (0.818) | -4.86 (0.797)
  Week 12 (n=150, 142, 148, 155) | 0.29 (0.883) | -4.08 (0.907) | -2.98 (0.887) | -4.65 (0.867)
  Week 16 (n=150, 142, 148, 155) | 0.26 (0.829) | -4.49 (0.852) | -3.65 (0.833) | -2.73 (0.814)
  Week 20 (n=150, 142, 148, 155) | -1.02 (0.844) | -4.56 (0.868) | -4.61 (0.848) | -3.06 (0.829)
  Week 26 (n=150, 142, 148, 155) | -0.47 (0.755) | -4.06 (0.776) | -3.86 (0.759) | -3.72 (0.742)

15. Secondary Outcome: Change From Baseline in Proinsulin/Insulin Ratio
Description: The ratio of proinsulin to insulin was calculated as proinsulin (pmol/L) / insulin (μIU/mL) at weeks 4, 8, 12, 16, 20 and 26 relative to the Baseline value. Least squares means were from an ANCOVA model with treatment and geographic region as class variables and Baseline proinsulin/insulin ratio as a covariate.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
ratio
  Week 4 (n=135, 133, 133, 145) | -0.073 (0.0150) | -0.047 (0.0151) | -0.080 (0.0151) | -0.056 (0.0144)
  Week 8 (n=149, 142, 146, 155) | -0.041 (0.0140) | -0.085 (0.0144) | -0.094 (0.0142) | -0.102 (0.0138)
  Week 12 (n=149, 142, 147, 155) | -0.062 (0.0122) | -0.098 (0.0125) | -0.123 (0.0123) | -0.095 (0.0120)
  Week 16 (n=149, 142, 147, 155) | -0.049 (0.0173) | -0.081 (0.0177) | -0.115 (0.0174) | -0.090 (0.0170)
  Week 20 (n=149, 142, 147, 155) | -0.057 (0.0173) | -0.076 (0.0177) | -0.124 (0.0174) | -0.119 (0.0169)
  Week 26 (n=149, 142, 147, 155) | -0.051 (0.0145) | -0.076 (0.0148) | -0.107 (0.0146) | -0.102 (0.0142)

16. Secondary Outcome: Change From Baseline in C-peptide Levels
Description: C-peptide is a byproduct created when the hormone insulin is produced and is measured by a blood test. Change from Baseline was assessed at Weeks 4, 8, 12, 16, 20 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline C-peptide as a covariate.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
ng/mL
  Week 4 (n=142, 141, 141, 146) | 0.057 (0.0740) | -0.551 (0.0741) | -0.593 (0.0741) | -0.452 (0.0729)
  Week 8 (n=158, 150, 153, 156) | 0.034 (0.0701) | -0.606 (0.0718) | -0.620 (0.0711) | -0.547 (0.0704)
  Week 12 (n=158, 150, 154, 156) | -0.040 (0.0676) | -0.612 (0.0693) | -0.534 (0.0684) | -0.536 (0.0680)
  Week 16 (n=158, 150, 154, 156) | 0.037 (0.0801) | -0.604 (0.0822) | -0.424 (0.0810) | -0.353 (0.0805)
  Week 20 (n=158, 150, 154, 156) | -0.097 (0.0783) | -0.623 (0.0803) | -0.556 (0.0792) | -0.374 (0.0787)
  Week 26 (n=158, 150, 154, 156) | -0.068 (0.0752) | -0.577 (0.0771) | -0.541 (0.0760) | -0.444 (0.0756)

17. Secondary Outcome: Change From Baseline in Calculated Homeostatic Model Assessment Insulin Resistance
Description: The Homeostasis Model Assessment of insulin resistance (HOMA IR) measures insulin resistance based on fasting glucose and insulin measurements:
  HOMA IR = fasting plasma insulin (µIU/mL) * fasting plasma glucose (mmol/L) / 22.5
  A higher number indicates a greater degree of insulin resistance. The change from Baseline in HOMA IR was assessed at Weeks 12 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline HOMA IR as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: insulin resistance
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
insulin resistance
  Week 12 (n=139, 132, 137, 143) | -0.814 (0.5309) | -3.479 (0.5458) | -2.905 (0.5348) | -3.877 (0.5236)
  Week 26 (n=145, 134, 144, 148) | -1.353 (0.3566) | -3.350 (0.3717) | -3.646 (0.3579) | -3.508 (0.3532)

18. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment Beta Cell Function
Description: The Homeostasis Model Assessment (HOMA) estimates steady state beta cell function (%B) as a percentage of a normal reference population.
  HOMA %B = 20 * insulin (µIU/mL) / fasting plasma glucose (mmol/L) - 3.5
  The change from Baseline in the homeostasis model assessment of beta cell function was assessed at Weeks 12 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline HOMA beta cell function as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage beta cell function
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
percentage beta cell function
  Week 12 (n= 139, 132, 137, 143) | 15.133 (4.2787) | 17.328 (4.3868) | 30.266 (4.3006) | 22.134 (4.2098)
  Week 26 (n=145, 134, 144, 148) | 10.472 (8.5306) | 17.500 (8.8718) | 39.153 (8.5455) | 24.887 (8.4285)

19. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from Baseline in body weight was assessed at Weeks 8, 12, 20 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and Baseline weight as a covariate.
Time Frame: Baseline and Weeks 8, 12, 20 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
kg
  Week 8 (n=155, 146, 152, 151) | -0.34 (0.184) | 0.58 (0.189) | 0.82 (0.185) | 0.70 (0.186)
  Week 12 (n=159, 147, 155, 154) | -0.78 (0.227) | 0.96 (0.236) | 1.35 (0.230) | 1.22 (0.230)
  Week 20 (n=159, 147, 155, 154) | -0.47 (0.265) | 1.56 (0.275) | 2.36 (0.268) | 1.86 (0.269)
  Week 26 (n=159, 147, 155, 154) | -0.29 (0.291) | 2.19 (0.302) | 3.14 (0.295) | 2.51 (0.296)

20. Secondary Outcome: Change From Baseline in Total Cholesterol Level
Description: Change from Baseline in total cholesterol level was assessed at Weeks 4, 8, 12, 16, 20 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline total cholesterol as a covariate.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
mg/dL
  Week 4 (n=146, 144, 142, 149) | -8.5 (2.22) | 0.9 (2.23) | -0.4 (2.25) | -5.3 (2.20)
  Week 8 (n=160, 151, 154, 158) | -5.4 (2.30) | 7.2 (2.37) | -0.3 (2.34) | -1.2 (2.31)
  Week 12 (n=160, 151, 155, 158) | -4.0 (2.43) | 4.9 (2.51) | -0.6 (2.47) | 4.4 (2.45)
  Week 16 (n=160, 151, 155, 158) | -4.3 (2.42) | 4.6 (2.49) | 3.8 (2.46) | 4.7 (2.44)
  Week 20 (n=160, 151, 155, 158) | -2.9 (2.67) | 4.5 (2.75) | -0.3 (2.71) | -0.6 (2.69)
  Week 26 (n=160, 151, 155, 158) | -0.5 (2.61) | 6.5 (2.68) | 3.7 (2.65) | 4.0 (2.62)

21. Secondary Outcome: Change From Baseline in Low-Density Lipoprotein Cholesterol
Description: Change from Baseline in low-density lipoprotein cholesterol (LDL-C) was assessed at Weeks 4, 8, 12, 16, 20 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline LDL cholesterol as a covariate.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
mg/dL
  Week 4 (n=137, 130, 135, 142) | -3.5 (1.88) | 2.8 (1.93) | 2.2 (1.89) | -2.8 (1.85)
  Week 8 (n=152, 139, 147, 153) | -0.5 (1.96) | 7.6 (2.05) | 2.6 (1.99) | 1.3 (1.95)
  Week 12 (n=154, 140, 148, 154) | 0.8 (2.02) | 5.8 (2.12) | 1.4 (2.06) | 3.9 (2.02)
  Week 16 (n=154, 140, 148, 154) | 1.8 (2.22) | 6.6 (2.33) | 5.3 (2.27) | 4.6 (2.22)
  Week 20 (n=154, 140, 148, 154) | 0.9 (2.27) | 7.4 (2.38) | 2.1 (2.32) | 0.5 (2.27)
  Week 26 (n=154, 140, 148, 154) | 2.0 (2.22) | 8.1 (2.33) | 4.6 (2.27) | 3.8 (2.22)

22. Secondary Outcome: Change From Baseline in High-Density Lipoprotein Cholesterol
Description: Change from Baseline in high-density lipoprotein cholesterol (HDL-C) was assessed at Weeks 4, 8, 12, 16, 20 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline HDL cholesterol as a covariate.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
mg/dL
  Week 4 (n=146, 144, 142, 149) | -0.2 (0.54) | 3.0 (0.54) | 3.8 (0.55) | 3.0 (0.54)
  Week 8 (n=160, 151, 154, 158) | 0.5 (0.56) | 4.7 (0.58) | 5.0 (0.57) | 4.8 (0.57)
  Week 12 (n=160, 151, 155, 158) | 0.9 (0.64) | 6.0 (0.66) | 6.4 (0.65) | 6.5 (0.65)
  Week 16 (n=160, 151, 155, 158) | 0.9 (0.57) | 5.2 (0.58) | 6.0 (0.58) | 5.9 (0.57)
  Week 20 (n=160, 151, 155, 158) | 0.5 (0.59) | 4.7 (0.60) | 5.6 (0.60) | 5.6 (0.59)
  Week 26 (n=160, 151, 155, 158) | 0.8 (0.64) | 5.7 (0.66) | 6.2 (0.65) | 6.2 (0.64)

23. Secondary Outcome: Change From Baseline in Triglyceride Levels
Description: Change from Baseline in triglycerides was assessed at Weeks 4, 8, 12, 16, 20 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline triglycerides as a covariate.
Time Frame: Baseline and Weeks 4, 8, 12, 16, 20 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
mg/dL
  Week 4 (n=146, 144, 142, 149) | -28.2 (8.60) | -43.2 (8.63) | -51.7 (8.70) | -32.1 (8.51)
  Week 8 (n=160, 151, 154, 158) | -34.8 (6.51) | -38.2 (6.69) | -61.6 (6.63) | -51.9 (6.56)
  Week 12 (n=160, 151, 155, 158) | -36.4 (6.90) | -47.9 (7.09) | -64.3 (7.00) | -45.4 (6.95)
  Week 16 (n=160, 151, 155, 158) | -44.5 (5.74) | -48.3 (5.90) | -54.6 (5.82) | -43.9 (5.78)
  Week 20 (n=160, 151, 155, 158) | -29.9 (7.35) | -46.6 (7.56) | -59.3 (7.46) | -46.5 (7.41)
  Week 26 (n=160, 151, 155, 158) | -24.7 (6.83) | -46.6 (7.02) | -56.2 (6.92) | -43.1 (6.88)

24. Secondary Outcome: Change From Baseline in Free Fatty Acids
Description: Change from Baseline in free fatty acids (FFA) was assessed at Weeks 12 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline free fatty acid as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
mmol/L
  Week 12 (n=148, 136, 140, 147) | -0.0404 (0.01643) | -0.0990 (0.01716) | -0.1061 (0.01690) | -0.0805 (0.01650)
  Week 26 (n=154, 136, 147, 150) | -0.0429 (0.01624) | -0.0680 (0.01729) | -0.0881 (0.01662) | -0.1013 (0.01647)

25. Secondary Outcome: Change From Baseline in Plasminogen Activator Inhibitor-1
Description: Change from Baseline in plasminogen activator inhibitor-1 was assessed at Weeks 12 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline plasminogen activator inhibitor-1 as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
ng/mL
  Week 12 (n=136, 127, 131, 133) | -1.58 (2.815) | -4.23 (2.909) | -9.63 (2.870) | -11.87 (2.849)
  Week 26 (n=145, 129, 142, 137) | 1.71 (3.151) | -5.45 (3.341) | -7.14 (3.189) | -8.38 (3.246)

26. Secondary Outcome: Change From Baseline in High-sensitivity C-Reactive Protein
Description: Change from Baseline in high-sensitivity C-Reactive Protein (hsCRP) was assessed at Weeks 12 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline hsCRP as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
mg/L
  Week 12 (n=147, 134, 138, 146) | -0.4497 (0.41497) | -1.7446 (0.43493) | -1.5346 (0.42831) | -2.2771 (0.41646)
  Week 26 (n=153, 135, 144, 149) | -0.1851 (0.42623) | -1.0391 (0.45388) | -1.9763 (0.43925) | -1.9796 (0.43182)

27. Secondary Outcome: Change From Baseline in Adiponectin
Description: Change from Baseline in adiponectin was assessed at Weeks 12 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline adiponectin as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: μg/mL
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
μg/mL
  Week 12 (n=148, 137, 141, 147) | -0.28 (0.560) | 6.35 (0.582) | 8.10 (0.575) | 7.50 (0.562)
  Week 26 (n=154, 137, 147, 149) | -0.09 (0.570) | 6.90 (0.605) | 6.85 (0.586) | 7.16 (0.581)

28. Secondary Outcome: Change From Baseline in Apolipoprotein A1
Description: Change from Baseline in Apolipoprotein A1 was assessed at Weeks 12 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and Baseline apolipoprotein A1 as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
mg/dL
  Week 12 (n=140, 138, 137, 144) | -1.6 (1.57) | 2.3 (1.58) | 1.0 (1.59) | 1.7 (1.55)
  Week 26 (n=149, 139, 146, 146) | -4.5 (1.59) | 1.2 (1.64) | 0.8 (1.60) | 1.6 (1.60)

29. Secondary Outcome: Change From Baseline in Apolipoprotein A2
Description: Change from Baseline in apolipoprotein A2 was assessed at Weeks 12 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline apolipoprotein A2 as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
mg/dL
  Week 12 (n=140, 138, 137, 144) | -0.1 (0.41) | 3.4 (0.41) | 2.8 (0.41) | 3.2 (0.40)
  Week 26 (n=149, 139, 146, 146) | -0.3 (0.41) | 2.9 (0.43) | 2.5 (0.42) | 2.6 (0.42)

30. Secondary Outcome: Change From Baseline in Apolipoprotein B
Description: Change from Baseline in apolipoprotein B was assessed at Weeks 12 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline apolipoprotein B as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
mg/dL
  Week 12 (n=140, 138, 137, 143) | -4.0 (1.76) | -5.0 (1.78) | -9.8 (1.78) | -5.9 (1.74)
  Week 26 (n=149, 139, 146, 146) | -2.5 (1.84) | -3.7 (1.91) | -7.9 (1.86) | -6.4 (1.86)

31. Secondary Outcome: Change From Baseline in Apolipoprotein C-III
Description: Change from Baseline in apolipoprotein C-III was assessed at Weeks 12 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline apolipoprotein C-III as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
mg/dL
  Week 12 (n=140, 138, 138, 144) | -0.5 (0.30) | -0.3 (0.30) | -0.8 (0.30) | -0.3 (0.30)
  Week 26 (n=149, 139, 147, 146) | -0.4 (0.28) | -0.2 (0.29) | -0.3 (0.28) | -0.4 (0.28)

32. Secondary Outcome: Change From Baseline in Nuclear Magnetic Resonance Lipid Fractionation Total Triglycerides
Description: Nuclear Magnetic Resonance (NMR) lipid fractionation was used to assess the change from Baseline in total triglyceride levels at Weeks 12 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline NMR total triglycerides as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 147 | 133 | 141 | 147
mg/dL
  Week 12 (n=139, 132, 132, 141) | -14.9 (6.36) | -25.0 (6.52) | -39.7 (6.52) | -23.7 (6.32)
  Week 26 (n=147, 133, 141, 147) | -7.6 (5.82) | -20.2 (6.11) | -28.8 (5.94) | -22.6 (5.82)

33. Secondary Outcome: Change From Baseline in Very Low Density Lipoprotein (VLDL) / Chylomicron Particles
Description: The change from Baseline in levels of total VLDL/chylomicron particles and large VLDL/chylomicron particles was assessed by NMR lipid fractionation at Weeks 12 and 26.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline VLDL/chylomicron particles as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
nmol/L
  Total Particles - Week 12 (n=139, 132, 132, 141) | -6.59 (2.600) | 0.70 (2.663) | -9.63 (2.664) | -2.67 (2.578)
  Total Particles - Week 26 (n=147, 133, 141, 147) | -4.97 (2.831) | 4.94 (2.976) | -0.73 (2.888) | -1.17 (2.828)
  Large Particles - Week 12 (n=139, 132, 132, 141) | -0.94 (0.511) | -1.83 (0.525) | -2.63 (0.525) | -2.06 (0.508)
  Large Particles - Week 26 (n=147, 133, 141, 147) | -0.18 (0.480) | -1.96 (0.505) | -2.37 (0.490) | -2.11 (0.480)

34. Secondary Outcome: Change From Baseline in VLDL / Chylomicron Triglycerides
Description: The change from Baseline in levels of VLDL/chylomicron triglycerides was assessed by NMR lipid fractionation at Weeks 12 and 26.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline VLDL/chylomicron triglycerides as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
mg/dL
  Week 12 (n=139, 132, 132, 141) | -14.4 (6.34) | -25.6 (6.50) | -39.5 (6.50) | -24.2 (6.30)
  Week 26 (n=147, 133, 141, 147) | -8.2 (5.79) | -22.0 (6.08) | -29.7 (5.90) | -23.3 (5.79)

35. Secondary Outcome: Change From Baseline in VLDL Particles
Description: The change from Baseline in levels of medium VLDL particles and small VLDL particles was assessed by NMR fractionation at Weeks 12 and 26.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline VLDL particles as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
nmol/L
  Medium Particles - Week 12 (n=139, 132, 132, 141) | -3.20 (1.639) | -2.30 (1.678) | -8.52 (1.679) | -4.69 (1.625)
  Medium Particles - Week 26 (n=147, 133, 141, 147) | -0.23 (1.784) | -0.39 (1.874) | -3.76 (1.819) | -3.58 (1.782)
  Small Particles - Week 12 (n=139, 132, 132, 141) | -1.74 (1.617) | 4.77 (1.662) | 1.18 (1.660) | 3.71 (1.607)
  Small Particles - Week 26 (n=147, 133, 141, 147) | -4.11 (1.710) | 7.16 (1.802) | 5.22 (1.746) | 4.36 (1.711)

36. Secondary Outcome: Change From Baseline in Mean VLDL Particle Size
Description: Change from Baseline in mean VLDL particle size was assessed by NMR lipid fractionation at Weeks 12 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline mean VLDL particle size as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
nm
  Week 12 (n=139, 132, 132, 141) | -0.97 (0.668) | -3.97 (0.688) | -2.92 (0.687) | -2.85 (0.665)
  Week 26 (n=147, 133, 141, 147) | 0.30 (0.607) | -3.71 (0.640) | -4.21 (0.620) | -2.80 (0.607)

37. Secondary Outcome: Change From Baseline in Intermediate Density Lipoprotein (IDL) Particles
Description: The change from Baseline in levels of IDL particles was assessed by NMR fractionation at Weeks 12 and 26.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline IDL particles as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
nmol/L
  Week 12 (n=139, 132, 132, 141) | -2.9 (3.63) | -1.0 (3.72) | -2.9 (3.73) | -4.0 (3.61)
  Week 26 (n=147, 133, 141, 147) | 0.5 (3.68) | 2.1 (3.86) | -1.0 (3.75) | -5.8 (3.68)

38. Secondary Outcome: Change From Baseline in Low Density Lipoprotein (LDL) Particles
Description: The change from Baseline in levels of total, large, medium-small, total small and very small LDL particles was assessed by NMR fractionation at Weeks 12 and 26.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline LDL particles as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nmol/L
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
nmol/L
  Total Particles - Week 12 (n=139, 132, 132, 141) | -11.9 (28.57) | -104.1 (29.34) | -207.0 (29.33) | -181.8 (28.40)
  Total Particles - Week 26 (n=147, 133, 141, 147) | 60.9 (30.67) | -75.6 (32.29) | -169.9 (31.31) | -177.1 (30.68)
  Large Particles - Week 12 (n=139, 132, 132, 141) | 15.3 (15.16) | 98.8 (15.52) | 129.4 (15.54) | 142.1 (15.05)
  Large Particles - Week 26 (n=147, 133, 141, 147) | 2.6 (15.32) | 120.4 (16.10) | 146.6 (15.63) | 155.5 (15.33)
  Medium-Small - Week 12 (n=139, 132, 132, 141) | -6.2 (6.25) | -41.4 (6.41) | -65.8 (6.41) | -65.8 (6.20)
  Medium-Small - Week 26 (n=147, 133, 141, 147) | 9.9 (6.42) | -40.1 (6.75) | -63.0 (6.55) | -66.6 (6.41)
  Total Small - Week 12 (n=139, 132, 132, 141) | -27.8 (31.91) | -200.3 (32.71) | -331.2 (32.73) | -320.0 (31.66)
  Total Small - Week 26 (n=147, 133, 141, 147) | 54.5 (33.34) | -195.8 (35.04) | -313.8 (34.01) | -327.4 (33.30)
  Very Small - Week 12 (n=139, 132, 132, 141) | -20.9 (26.22) | -159.2 (26.88) | -265.7 (26.90) | -254.2 (26.02)
  Very Small - Week 26 (n=147, 133, 141, 147) | 45.1 (27.44) | -156.0 (28.83) | -250.9 (27.98) | -260.8 (27.40)

39. Secondary Outcome: Change From Baseline in Mean LDL Particle Size
Description: Change from Baseline in mean LDL particle size was assessed by NMR lipid fractionation at Weeks 12 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline mean LDL particle size as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
nm
  Week 12 (n=139, 132, 132, 141) | 0.09 (0.051) | 0.44 (0.053) | 0.63 (0.053) | 0.58 (0.051)
  Week 26 (n=147, 133, 141, 147) | -0.02 (0.052) | 0.44 (0.054) | 0.65 (0.053) | 0.61 (0.052)

40. Secondary Outcome: Change From Baseline in High Density Lipoprotein (HDL) Particles
Description: The change from Baseline in levels of total, large, medium and small HDL particles was assessed by NMR fractionation at Weeks 12 and 26.
  Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline HDL particles as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: µmol/L
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
µmol/L
  Total Particles - Week 12 (n=139, 132, 132, 141) | 0.18 (0.350) | 0.92 (0.359) | 0.11 (0.359) | 0.54 (0.348)
  Total Particles - Week 26 (n=147, 133, 141, 147) | 0.81 (0.359) | 1.67 (0.377) | 1.01 (0.367) | 1.03 (0.359)
  Large Particles - Week 12 (n=139, 132, 132, 141) | 0.07 (0.195) | 0.99 (0.200) | 0.98 (0.200) | 1.31 (0.193)
  Large Particles - Week 26 (n=147, 133, 141, 147) | -0.06 (0.197) | 1.14 (0.207) | 1.24 (0.201) | 1.31 (0.197)
  Medium Particles - Week 12 (n=139, 132, 132, 141) | -0.26 (0.311) | 0.72 (0.319) | 1.60 (0.320) | 1.61 (0.308)
  Medium Particles - Week 26 (n=147, 133, 141, 147) | -0.26 (0.313) | 0.95 (0.329) | 1.19 (0.320) | 1.30 (0.312)
  Small Particles - Week 12 (n=139, 132, 132, 141) | 0.50 (0.412) | -0.68 (0.423) | -2.65 (0.423) | -2.42 (0.410)
  Small Particles - Week 26 (n=147, 133, 141, 147) | 1.24 (0.412) | -0.28 (0.433) | -1.58 (0.421) | -1.63 (0.413)

41. Secondary Outcome: Change From Baseline in Mean HDL Particle Size
Description: Change from Baseline in mean HDL particle size was assessed by NMR lipid fractionation at Weeks 12 and 26. Least squares means are from an ANCOVA model with treatment and geographic region as class variables and baseline mean HDL particle size as a covariate.
Time Frame: Baseline and Weeks 12 and 26.
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: nm
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Number analyzed (Participants) | 164 | 163 | 164 | 163
nm
  Week 12 (n=139, 132, 132, 141) | -0.02 (0.024) | 0.09 (0.025) | 0.17 (0.025) | 0.15 (0.024)
  Week 26 (n=147, 133, 141, 147) | -0.03 (0.024) | 0.08 (0.025) | 0.15 (0.024) | 0.14 (0.024)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent until the end of the study, and from spontaneous reporting for 30 days after the end of treatment.
Description: At each study visit, the investigator assessed whether any events had occurred. Patients could report events at any other time during the study. All events, whether reported by the patient or observed by the investigator, were documented, whether or not the investigator concluded the event to be related to the drug treatment.
Arm/Group | Alogliptin 25 mg | Pioglitazone 30 mg | Alogliptin 25 mg + Pioglitazone 30 mg | Alogliptin 12.5 mg + Pioglitazone 30 mg
Serious Adverse Events (participants affected / at risk) | 1/164 | 6/163 | 8/164 | 1/163
Other Adverse Events (participants affected / at risk) | 19/164 | 25/163 | 37/164 | 24/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 25 mg (N=164) | Pioglitazone 30 mg (N=163) | Alogliptin 25 mg + Pioglitazone 30 mg (N=164) | Alogliptin 12.5 mg + Pioglitazone 30 mg (N=163)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Cervicitis (Infections and infestations) | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 25 mg (N=164) | Pioglitazone 30 mg (N=163) | Alogliptin 25 mg + Pioglitazone 30 mg (N=164) | Alogliptin 12.5 mg + Pioglitazone 30 mg (N=163)
Headache (Nervous system disorders) | 11 | 11 | 20 | 14
Urinary tract infection (Infections and infestations) | 5 | 4 | 9 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 10 | 3
Oedema peripheral (General disorders) | 2 | 9 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.